CLINICAL TRIAL: NCT03199326
Title: Collaborative Care for Infants at Risk
Acronym: CCIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Kristine Campbell, Associate Professor, Pediatrics, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00098047
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Child Abuse; Primary Health Care; Child Welfare

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Surveys will be collected without knowledge of intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care (Experimental): CPS caseworkers will be randomized to collaborative or comparison practice. For any infant investigated by a caseworker in the collaborative practice, the caseworkers will conduct a standard CPS investigation. Additionally, caseworkers will seek parental permission to contact an identified primary health care provider at two points in the CPS investigation for information sharing related to health needs, social risks, and recommended interventions.
  Interventions: Other: Collaborative Care
- Comparison Care (No Intervention): CPS caseworkers will be randomized to collaborative or comparison practice. For any infant investigated by a caseworker in the comparison practice, the caseworkers will conduct a standard CPS investigation.

INTERVENTIONS:
Other: Collaborative Care — CPS caseworkers will explain collaborative care to parents, ask parents to allow communication with an infant's primary care provider, and have willing parents sign a release allowing communication with the infant's provider during the investigation. Caseworkers will make at least two attempts to contact identified providers with parental consent. In the first week, caseworkers will contact the provider, identify the infant, and summarize the child maltreatment concerns. The caseworker will ask whether the provider recognizes any additional strengths or vulnerabilities for the infant. Prior to case closure, caseworkers will provide a summary of investigation findings, disposition, and service referrals including placement changes, safety planning, family preservation, and community resources, with a summary letter delivered to the provider after case closure.
  Arms: Collaborative Care

SUMMARY:
This study evaluates the feasibility, acceptability, and impact of a collaborative care practice for infants investigated by state Child Protective Services (CPS) for suspected maltreatment. Recognizing the vulnerability of infants referred into CPS in the first year of life, as well as the frequent contact of infants with health care providers in the first year of life, the investigators will conduct a RCT to measure the impact of a collaborative practice model linking CPS caseworkers with primary health care providers during an investigation for suspected infant maltreatment. With this trial, the investigators will ask (3a) Can a collaborative practice model improve parent-reported infant health-related quality of life 6 months following child welfare involvement for suspected infant maltreatment? and (3b) Does a collaborative practice model impact repeat child welfare involvement for suspected child maltreatment over 6 months?

ELIGIBILITY:
Inclusion Criteria:

* Less than 12 months of age at referral
* Involved in a child welfare investigation for suspected maltreatment
* Investigation occurring in Utah DCFS Salt Lake Valley or Western regions

Exclusion Criteria:

For the primary and selected secondary outcomes,

* Caregiver with primary spoken language other than English or Spanish,
* CPS caseworkers not yet randomized to a practice arm
* Infants in out-of-home placement at the time of referral or case closure,
* Infants suffering fatal maltreatment
* Prior investigation of an infant in a household during study timeframe (e.g., twins, infant siblings, and repeat referrals will be excluded).

For other secondary outcomes related to CPS outcomes, language exclusion will not be considered.

Ages: 0 Days to 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 468 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Infant Health Related Quality of Life | Change from baseline to 6 months following CPS case closure
  Difference in Change in Infant Health Related Quality of Life based on practice arm

SECONDARY OUTCOMES:
Parent Perception of Child Welfare and Child Health Care | at baseline (child welfare) and at 6 months (child health care)
  Difference in parent perceptions of child welfare and child health care based on practice arm
Repeat Child Welfare Involvement | 6 months after CPS case closure
  Repeat Child Welfare Involvement

OTHER OUTCOMES:
Engagement of child welfare caseworkers | baseline
  Proportion of eligible cases investigated that were offered collaborative practice
Acceptance of parents | baseline
  Proportion of cases offered collaborative practice in which parents allowed practice
Recruiting and retention of high-risk longitudinal cohort | baseline and 6 months
  Proportion of eligible cases willing to enroll in and follow-up with researchers

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Campbell, MD, MSc, Principal Investigator — University of Utah
Locations (1):
- The Center for Safe and Healthy Families, Primary Children's Hospital Eccles Outpatient Building, 81 North Mario Capecchi Dr 4E-200, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No